CLINICAL TRIAL: NCT04551833
Title: Tramadol Versus Dexamethasone as Adjuvant to Levobupivacaine Under Ultrasound Guided Supraclavicular Block of Forearm Fractures
Brief Title: Tramadol Versus Dexamethasone as Adjuvant to Levobupivacaine Supraclavicular Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Gamal, Resident of Anesthesia, ICU and Pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: supraclavicular block
Record Dates: First submitted 2020-03-18; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Regional Anesthesia
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (T) : 30 patients (Tramadol group) (Experimental): Patient will receive 0.4 mL/kg of 0.5% Levobupivacaine plus 1.5 mg/kg Tramadol.
  Interventions: Drug: Levobupivacaine
- Group (D) : 30 patients (Dexamethasone group): (Experimental): Patient will receive 0.4 mL/kg of 0.5% Levobupivacaine plus 8mg of Dexamethasone
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — Tramadol versus Dexamethasone as adjuvant to Levobupvacain

SUMMARY:
The investigator's aim will be to compare the efficacy of perineural tramadol and dexamethasone added to levobupivacaine in prolonging postoperative analgesia in patient undergoing open reduction and internal fixation for forearm fractures.

Primary outcome: duration of postoperative analgesia. Secondary outcome: include [The anesthesia onset time, total rescue analgesic consumption in the 1st 24-hour and the presence of complications and side effects.

DETAILED DESCRIPTION:
Strategies to prolong brachial plexus nerve blocks analgesia beyond the pharmacological duration of the local anaesthetic used include placement of indwelling perineural catheters to allow prolonged infusion or the co-administration of adjuvants such as epinephrine, alpha 2 agonists (as clonidine and dexmedetomidine), midazolam, or the corticosteroid dexamethasone .

Dexamethasone improves the quality and duration of peripheral nerve block over local anaesthetic alone. This is thought to be mediated by attenuating the release of inflammatory mediators, reducing ectopic neuronal discharge, and inhibiting potassium channel-mediated discharge of nociceptive C-fibres .

Tramadol is a unique opioid with two modes of action for inhibition of pain, an opioid action mediated by the μ receptor and a non-opioid action mediated by α-2-adrenergic and serotoninergic activity .The monoaminergic activity of tramadol inhibits the descending pain pathways, resulting in suppression of nociceptive transmission at the spinal level . Tramadol also exhibits local anaesthetic properties by blocking K+ channels .Many studies have characterized the effects of tramadol as an adjuvant to local anaesthetic in brachial plexus block .

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status I-II patients older than 18years and scheduled for internal fixation for forearm fractures
* Both sexes

Exclusion Criteria:

* Patients with known allergy to the study drugs
* Skin infection at site of needle puncture
* Significant organ dysfunction
* Coagulopathy
* Drug or alcohol abuse
* Epilepsy and psychiatric illness that would interfere with perception and assessment of pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Duration of postoperative analgesia in hours | 24 hours
  Duration of postoperative analgesia in hours

SECONDARY OUTCOMES:
The anesthesia onset time | 20 minutes
  Anasthesia onset
Dose of Paracetamol as rescue analgesia in mg | 24 hours
  Rescue Analgesia in mg
Presence of complications and side effects | 24 hours
  complications and side effects

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao WL, Ou XF, Liu J, Zhang WS. Perineural versus intravenous dexamethasone as an adjuvant in regional anesthesia: a systematic review and meta-analysis. J Pain Res. 2017 Jul 4;10:1529-1543. doi: 10.2147/JPR.S138212. eCollection 2017. PMID 28740419
- [Background] Pehora C, Pearson AM, Kaushal A, Crawford MW, Johnston B. Dexamethasone as an adjuvant to peripheral nerve block. Cochrane Database Syst Rev. 2017 Nov 9;11(11):CD011770. doi: 10.1002/14651858.CD011770.pub2. PMID 29121400
- [Background] Nagpal V, Rana S, Singh J, Chaudhary SK. Comparative study of systemically and perineurally administered tramadol as an adjunct for supraclavicular brachial plexus block. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):191-5. doi: 10.4103/0970-9185.155147. PMID 25948899